CLINICAL TRIAL: NCT06157827
Title: An Open-label, Multicenter Phase Ib/II Clinical Study to Evaluate the Safety and Efficacy of LBL-024 Combined With Etoposide and Platinum in the First-line Treatment of Patients With Advanced Neuroendocrine Carcinoma (NEC)
Brief Title: A Clinical Trial of LBL-024 Combined With Etoposide and Platinum in Patients With Advanced Neuroendocrine Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBL-024-CN002
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Advanced Neuroendocrine Carcinoma
MeSH Terms: interventions — Injections; Etoposide; Carboplatin; atezolizumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBL-024+Etoposide+Carboplatin/Cisplatin (Experimental): LBL-024+Etoposide+Carboplatin/Cisplatin Injection，dose A、dose B or dose C; Q3W
  Interventions: Drug: LBL-024 for Injection; Drug: Etoposide Injection; Drug: Carboplatin Injection; Drug: Cisplatin injection
- Atezolizumab+Etoposide+Carboplatin (Experimental): Atezolizumab+Etoposide+Carboplatin Injection，dose A ; Q3W
  Interventions: Drug: Etoposide Injection; Drug: Carboplatin Injection; Drug: Atezolizumab injection

INTERVENTIONS:
Drug: LBL-024 for Injection — Initial dose-MTD; Q3W; intravenous infusion
  Other Names: LBL-024
  Arms: LBL-024+Etoposide+Carboplatin/Cisplatin
Drug: Etoposide Injection — Initial dose（Dose was decided by the investigator according to the subject's condition）; Q3W; intravenous infusion
  Other Names: Etoposide
Drug: Carboplatin Injection — Initial dose（Dose was decided by the investigator according to the subject's condition）; Q3W; intravenous infusion
  Other Names: Carboplatin
Drug: Atezolizumab injection — Initial dose; Q3W; intravenous infusion
  Other Names: Atezolizumab
  Arms: Atezolizumab+Etoposide+Carboplatin
Drug: Cisplatin injection — Initial dose（Dose was decided by the investigator according to the subject's condition）; Q3W; intravenous infusion
  Other Names: Cisplatin
  Arms: LBL-024+Etoposide+Carboplatin/Cisplatin

SUMMARY:
An open-label, multicenter phase Ib/II clinical study to evaluate the safety and efficacy of LBL-024 combined with etoposide and platinum in the first-line treatment of patients with advanced neuroendocrine carcinoma (NEC)

DETAILED DESCRIPTION:
This trial includes two parts: phase Ib and phase II study. Phase Ib is a dose-escalation and Phase II is the dose optimization and dose expansion .

Phase Ib program to enroll patients with advanced neuroendocrine carcinoma (NEC) without systemic therapy.To sequentially evaluate the safety and tolerability of LBL-024 in combination with etoposide and platinum (cisplatin or carboplatin) at different doses by the dose-escalation method.

Phase II includes two stages, dose optimization and dose expansion.

The dose optimization part will conduct combination of LBL-024, which is a further optimization study in two dose groups, enrolling patients with EP-NEC who have not received systemic treatment, to fully assess the dose-exposure-effect relationship, and in combination with the target binding characteristics of LBL-024, pharmacokinetic/pharmacodynamic, efficacy and/or safety profile, considering multiple dimensions,To confirm the rationale for the recommended Phase 2 dose (RP2D).

The recommended Phase 2 dose (RP2D) will be determined based on the safety, tolerability, efficacy and PK data from the clinical studies of LBL-024.After obtaining the RP2D, a dose expansion study of combination dosing at the RP2D will be conducted to obtain adequate efficacy data.

This trial will enroll 178 patients in Phase Ib and Phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily agreed to participate by giving written informed consent for the trial，and Consent to follow trial treatment and visit schedule
2. aged 18-75 years (including borderline values) at the time of signing the informed consent form
3. Have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale
4. Have a life expectancy of at least 12 weeks
5. Subject has at least one measurable target lesion by RECIST 1.1 criteria
6. Fertile men and women of childbearing age are willing to take effective contraceptive measures (including abstinence, intrauterine devices, hormonal contraception, and correct use of condoms) from the signing of the informed consent form to 6 months after the last dose of the investigational drug; women of childbearing age include premenopausal women and women who had menopause less than two years ago. Blood pregnancy test results must be negative for women of childbearing age within 7 days prior to the initial dose of the investigational drug.

Exclusion Criteria:

1. Subjects who underwent major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the initial use of the investigational drug, or require elective surgery during the trial period
2. Use of immunomodulatory drugs within 14 days prior to the initial use of the investigational drug, including but not limited to thymosin, interleukin, and interferon
3. Systemic use of corticosteroidsor other immunosuppressants within 14 days prior to the initial use of the investigational drug;The following conditions are excluded: Treatment with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; short-term use of glucocorticoids for preventive therapy (e.g., to prevent contrast allergy)
4. Subjects with an active infection that currently requires intravenous anti infective therapy
5. History of immunodeficiency, including positive HIV antibody test results
6. Pregnant or lactating women
7. The investigator's assessment that there may be other factors affecting compliance among participants or that some may not be suitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy).
  ORR (including the rates of complete response (CR) and partial response (PR)), evaluated based on the RECIST 1.1, refers to the percentage of study subjects who achieve a complete response or partial response. It was used to evaluate the efficacy in Phase II .
Dose-limiting toxicities（DLT） | Within 3 weeks after receiving the first dose of the test drug (DLT assessment for subjects in dose escalation phase).
  DLT describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment. It was used to evaluate the safety in Phase Ib.
Maximum tolerated dose (MTD) | Within 3 weeks after receiving the first dose of the test drug (MTD assessment for subjects in dose escalation phase).
  MTD is defined as the hightest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first cycles. It was used to evaluate the tolerability in Phase Ib .
Progression-Free Survival(PFS) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy).
  PFS is defined as the time from randomization to disease progression or death from any cause.It was used to evaluate the efficacy in Phase II .

SECONDARY OUTCOMES:
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy
  Maximum serum concentration
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy
  After taking a single dose, Time to reach maximum plasma concentration
immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects
Duration of Response(DOR） | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy
  The period from the participants first achieving CR or PR to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: lin shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (24):
- China (24):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Anhui Cancer Hospital, Hefei, Anhui
  - Beijing GoBroad Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No